CLINICAL TRIAL: NCT02260323
Title: Compliance of Traditional Chinese Medicine in Young Patients With Rheumatic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Ph.D, Chengdu PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CT20141003
Record Dates: First submitted 2014-10-02; First posted 2014-10-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Chronic Rheumatic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patient-tailored anti-arthritis herbs (Experimental): patient use tailored anti-arthritis herbs
  Interventions: Other: patient-tailored anti-arthritis herbs
- patient-tailored DMARDs (Active Comparator): Patients use tailored DMARDs
  Interventions: Other: patient-tailored DMARDs

INTERVENTIONS:
Other: patient-tailored anti-arthritis herbs — patient use tailored anti-arthritis herbs
  Arms: patient-tailored anti-arthritis herbs
Other: patient-tailored DMARDs — patient use tailored disease-modifying antirheumatic drugs
  Other Names: patient-tailored disease-modifying antirheumatic drugs
  Arms: patient-tailored DMARDs

SUMMARY:
To evaluate the compliance of traditional Chinese medicine (TCM) in young people with Chronic rheumatic disease

ELIGIBILITY:
Inclusion Criteria:

* were between 18 and 35 years of age
* without use of TCM in the previous 3 months
* and had a Steinbrocker functional status of class I, II, or III

Exclusion Criteria:

* previous general health conditions disallowed their use of TCM
* were pregnant
* lack of motivation, remote from home, time-consuming,intervention, or other personal difficulties

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in HBCS(Hill-Bone Compliance Scale) score at 48 weeks | at 0 week, 12 weeks, 24 weeks, 48 weeks
Changes from baseline in MARS(Medication Adherence Rating Scale) score at 48 weeks | at 0 week, 12 weeks, 24 weeks, 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Chengdu Military Area Command PLA, Chengdu, Sichuan, China